CLINICAL TRIAL: NCT02473809
Title: The Effect of Liraglutide on Bone Turnover, Bone Mass and Bone Cell Function
Acronym: LIRABONE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07052015
Record Dates: First submitted 2015-06-08; First posted 2015-06-17 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Complications; Osteoporosis
MeSH Terms: conditions — Diabetes Complications; Osteoporosis | interventions — Liraglutide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Experimental): Liraglutide ("Victoza"), subcutaneous 1,8 mg once daily for 180 days
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): Saline, subcutaneous once daily for 180 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — Once daily
  Other Names: Victoza
  Arms: Liraglutide
Drug: Placebo — Once daily
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to test whether liraglutide, a drug approved and widely used in the treatment of type 2 diabetes, has an effect on bone mass and bone cell function. Type 2 diabetes may cause multiple complications, and it is well known that patients with type 2 diabetes have a higher risk of fractures. If Liraglutide can be demonstrated to have a positive effect on bone, this may be one among other factors to consider before the decision about specific treatment of type 2 diabetes is made for the individual patient.

DETAILED DESCRIPTION:
Background: Type 2 diabetes may cause complications such as ischemic heart disease, nephropathy, neuropathy, and retinopathy. Several epidemiologic and animal studies also suggest that fracture risk is increased in diabetes.

Bone is remodelled throughout life through bone resorption by the bone resorbing cells, the osteoclasts, and by bone formation by the bone forming cells, the osteoblasts. Bone remodelling can be monitored by biochemical markers of bone turnover and the effect of bone remodelling can be measured by changes in bone mineral density (BMD) by Dual X-ray absorptiometry (DXA) or bone structure by quantitative CT (QCT) or high resolution peripheral QCT (HRpQCT). The remodelling activity and the balance between resorption and formation are influenced by many factors including food consumption. The gut hormone glucagon-like polypeptide 1 (GLP-1) is released in relation to food intake and reduces serum levels of glucagon, increases serum levels of insulin, and reduces blood glucose in diabetes. Liraglutide is a GLP-1 analogue and has been approved for the treatment of type 2 diabetes.

Aim: To investigate the effect of the GLP-1 analogue Liraglutide on bone turnover, bone mass, and bone structure in patients with type 2 diabetes.

Methods: The clinical study will be conducted as a randomised, double-blinded, placebo-controlled, prospective, clinical trial with comparative treatment regimes with either subcutaneous Liraglutide or subcutaneous placebo injections.

Perspectives: The project will bring new knowledge about the possible effects of GLP-1 analogues on bone turnover and structure. This is important given that type 2 diabetes deteriorates bone health and increases risk of fractures. If Liraglutide can be demonstrated to have a positive effect on bone, this may be one among other factors to consider before the decision about specific treatment of type 2 diabetes is made for the individual patient.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Diagnosis of type 2 diabetes (HbA1c > 48 mmol/mol)
* Age older than 30 years

Exclusion Criteria:

* Type 1 diabetes
* Treatment with insulin
* Body weight > 140 kg
* HbA1c > 75 mmol/mol
* Treatment with GLP-1 analogues, Dipeptidyl peptidase-4 inhibitors, or glitazones
* Chronic kidney disease
* Hepatic disease
* Pancreatitis
* Inflammatory bowel disease
* Osteoporosis
* Family or personal history of medullary thyroid carcinoma
* Treatment with glucocorticoids
* Hormone replacement therapy
* Diabetic gastroparesis
* Pregnancy or lactation

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in collagen I cross-linked C-terminal telopeptide measured in serum | Days 0, 7, 28, 90, 180
  Collagen I cross-linked C-terminal telopeptide has been chosen as primary endpoint as the expected mechanism of action is reduction in bone resorption, and as it is the most responsive bone resorption marker.

SECONDARY OUTCOMES:
Change in bone alkaline phosphatase measured in serum | Days 0, 7, 28, 90, 180
Change in BMD evaluated by DXA | Days 0, 90, 180
Change in bone structure evaluated by QCT and HRpQCT | Days 0, 90, 180
Change in HbA1c | Days 0, 180
Change in osteocalcin measured in serum | Days 0, 7, 28, 90, 180
Change in procollagen type I N-terminal propeptide measured in serum | Days 0, 7, 28, 90, 180

CONTACTS AND LOCATIONS:
Overall Officials: Bente L Langdahl, MD PhD DMSc, Study Director — Department of Endocrinology and Internal Medicine, Aarhus University Hospital, Denmark
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus University Hospital, Aarhus, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fehmann HC, Hering BJ, Wolf MJ, Brandhorst H, Brandhorst D, Bretzel RG, Federlin K, Goke B. The effects of glucagon-like peptide-I (GLP-I) on hormone secretion from isolated human pancreatic islets. Pancreas. 1995 Aug;11(2):196-200. doi: 10.1097/00006676-199508000-00014. PMID 7479679
- [Background] Leslie WD, Rubin MR, Schwartz AV, Kanis JA. Type 2 diabetes and bone. J Bone Miner Res. 2012 Nov;27(11):2231-7. doi: 10.1002/jbmr.1759. Epub 2012 Sep 28. PMID 23023946
- [Background] Schwartz AV, Sellmeyer DE. Diabetes, fracture, and bone fragility. Curr Osteoporos Rep. 2007 Sep;5(3):105-11. doi: 10.1007/s11914-007-0025-x. PMID 17925191
- [Background] Vestergaard P. Discrepancies in bone mineral density and fracture risk in patients with type 1 and type 2 diabetes--a meta-analysis. Osteoporos Int. 2007 Apr;18(4):427-44. doi: 10.1007/s00198-006-0253-4. Epub 2006 Oct 27. PMID 17068657
- [Background] Yamada C, Yamada Y, Tsukiyama K, Yamada K, Udagawa N, Takahashi N, Tanaka K, Drucker DJ, Seino Y, Inagaki N. The murine glucagon-like peptide-1 receptor is essential for control of bone resorption. Endocrinology. 2008 Feb;149(2):574-9. doi: 10.1210/en.2007-1292. Epub 2007 Nov 26. PMID 18039776
- [Background] Nuche-Berenguer B, Lozano D, Gutierrez-Rojas I, Moreno P, Marinoso ML, Esbrit P, Villanueva-Penacarrillo ML. GLP-1 and exendin-4 can reverse hyperlipidic-related osteopenia. J Endocrinol. 2011 May;209(2):203-10. doi: 10.1530/JOE-11-0015. Epub 2011 Mar 3. PMID 21372151
- [Background] Su B, Sheng H, Zhang M, Bu L, Yang P, Li L, Li F, Sheng C, Han Y, Qu S, Wang J. Risk of bone fractures associated with glucagon-like peptide-1 receptor agonists' treatment: a meta-analysis of randomized controlled trials. Endocrine. 2015 Feb;48(1):107-15. doi: 10.1007/s12020-014-0361-4. Epub 2014 Jul 30. PMID 25074632